CLINICAL TRIAL: NCT06501534
Title: A Randomized, Open Label, Multicenter, Parallel-group, Positive-controlled, Dose Finding, and Phase II Study to Assess Efficacy and Safety of IBI128 in Chinese Gout Subjects
Brief Title: A Dose Finding Study to Assess Efficacy and Safety of IBI128 in Chinese Gout Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI128A201
Record Dates: First submitted 2024-07-02; First posted 2024-07-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Febuxostat 40mg (Active Comparator): Tablets, Once a day (QD), Per oral
  Interventions: Drug: Febuxostat
- IBI128 50mg (Experimental): Tablets, Once a day (QD), Per oral
  Interventions: Drug: IBI128
- IBI128 200mg (Experimental): Tablets, Once a day (QD), Per oral
  Interventions: Drug: IBI128
- IBI128 100mg (Experimental): Tablets, Once a day (QD), Per oral
  Interventions: Drug: IBI128

INTERVENTIONS:
Drug: Febuxostat — Tablets, Once a day (QD), Per oral
  Arms: Febuxostat 40mg
Drug: IBI128 — Other Names: LC350189, Tigulixostat,Tablets, Once a day (QD), Per oral
  Arms: IBI128 100mg; IBI128 200mg; IBI128 50mg

SUMMARY:
IBI128 (Tigulixostat) is a novel non-purine selective inhibitor of xanthine oxidase (XO). The XO inhibitors lower uric acid concentrations in serum by inhibiting the production of uric acid.

This ia a randomized, open label, multicenter, parallel-group, positive-controlled, dose finding, and Phase II study to assess efficacy and safety of IBI128 in chinese gout subjects.

ELIGIBILITY:
Inclusion criteria:

1. Participants must be aged between 18 and 75 years old (inclusive, as of the time of signing the informed consent form), with no gender restrictions;
2. Body Mass Index (BMI) should fall within the range of 18.0 to 40.0 kg/m² (including both ends of the range);
3. Subjects must meet the 2015 ACR/EULAR classification criteria for the diagnosis of gout (refer to Appendix 4);
4. At the screening stage, subjects must have a blood uric acid level of ≥480 μmol/L;
5. Subjects must voluntarily sign the informed consent form and agree to strictly adhere to the requirements outlined in this protocol.

Exclusion criteria (brief):

1. History of allergy to any component of Tigulixostat;
2. Previous allergy or intolerance to Febuxostat;
3. Subjects who have taken uric acid lowering medications within 2 weeks prior to screening;
4. Subjects who experienced an acute gout flare-up within 4 weeks prior to screening or immediately before the first dose administration;
5. Subjects considered to have secondary gout (elevated serum uric acid due to causes other than renal insufficiency);
6. Subjects with a history of xanthinuria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects in each treatment group with serum uric acid levels <360 μmol/L after continuous treatment for 16 weeks | Week 16

SECONDARY OUTCOMES:
The proportion of subjects in each treatment group with serum uric acid levels <300 μmol/L after continuous treatment for 16 weeks | Week 16
The proportion of subjects in each treatment group with serum uric acid levels <360, <300 μmol/L after continuous treatment for 2, 4, 8, 12 weeks | Week 2, 4, 8, 12
Absolute and percentage Changes in serum uric acid levels from baseline in subjects of each treatment group after continuous treatment for 2, 4, 8, 12, and 16 weeks | Baseline, Week 2, 4, 8, 12
The proportion of subjects experiencing gout flares and the number of gout flare occurrences within every 4 weeks from the first dose, among those receiving various doses of Tigulixostat tablets and Febuxostat tablets | Baseline through Week 16/18
Number of subjects with Adverse Event, Serious Adverse Events, Treatment Emergent Adverse Event, Adverse event of special interest | Baseline through Week 18/20
Number of subjects with clinically significant changes in physical examination results | Baseline through Week 16/18
  Clinically significant abnormal physical examination findings reported by the investigator.
Number of subjects with clinically significant changes in in vital sign | Baseline through Week 16/18
  Vital signs including body temperature, pulse, respiratory rate, SpO2 and blood pressure.
Number of subjects with clinically significant changes in clinical laboratory parameters | Baseline through Week 16/18
  Clinical laboratory parameters including white blood cell, red blood cell, hemoglobin, platelet, total cholesterol, triglyceride, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, serum creatinine, fasting serum glucose, toal bilirubin, direct bilirubin, alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase, alkaline phosphatase, serum potassium, creatine phosphokinase, hs-CRP, prothrombin time, thrombin time, activated partial thromboplastin time, international normalized ratio
Number of subjects with clinically significant changes in electrodiagram | Baseline through Week 16/18
  Electrodiagram parameters including PRinterval, heart rate, RRinterval, corrected QT interval by Fridericia's formula
Plasma concentration of Tigulixostat | Baseline through Week 16/18

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Fudan University HuaShan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No